CLINICAL TRIAL: NCT03467373
Title: A Phase Ib Study Evaluating Glofitamab (RO7082859) in Combination With Rituximab (R) or Obinutuzumab (G) Plus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (CHOP), or Polatuzumab Vedotin (POLA) Plus Rituximab (R), Cyclophosphamide, Doxorubicin, and Prednisone (CHP) in Participants With Relapsed or Refractory Non-Hodgkin Lymphoma (R/R NHL) or in Participants With Untreated Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: A Study of Glofitamab in Combination With Rituximab or Obinutuzumab Plus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (CHOP), or Polatuzumab Vedotin Plus Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone (CHP) in Participants With Non-Hodgkin Lymphomas or With DLBCL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP40126; 2017-003648-18 (EudraCT Number)
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: B-Cell Lymphoma; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin | interventions — glofitamab; obinutuzumab; Rituximab; tocilizumab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; polatuzumab vedotin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose Escalation r/r NHL (Experimental): Dose finding in participants with r/r NHL: the study will explore different doses of glofitamab in the induction period, starting at a dose of 70 mcg administered in combination with standard of care doses of G/R CHOP and R-CHOP every 3 weeks (Q3W). Participants with r/r NHL will receive 6 cycles of induction treatment (G/R-CHOP). Glofitamab will be administered using step-up dosing for Cycle 2 on Days 8 and 15, followed by single doses on Day 8 for Cycles 3-6. Participants who achieve a complete response (CR), partial response (PR), or stable disease (SD) at the end of induction (EOInd) may optionally receive post-induction treatment (referred to as maintenance) with glofitamab alone.
  The use of G versus R in Cycle 1 will be compared in parallel dose escalation cohorts.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab (G); Drug: Rituximab (R); Drug: Tocilizumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone
- Part 2: DLBCL G/R-CHOP (Experimental): Participants with untreated DLBCL will receive G-CHOP or R-CHOP in Cycle 1, followed by G/R-CHOP + glofitamab for subsequent cycles. Glofitamab will be administered using step-up dosing for Cycle 2 on Days 8 and 15, followed by single doses on Day 8 for Cycles 3-6 (up to 8). The starting dose of glofitamab for each arm may be one or more levels below the MTD/OBD determined in Part I.
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab (G); Drug: Rituximab (R); Drug: Tocilizumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone
- Part 2: DLBCL Pola-R-CHP (Experimental): Participants with untreated DLBCL will receive Pola-R-CHP + glofitamab on Day 1 of each 21-day cycle for a maximum of 6 cycles. Glofitamab will be administered using step-up dosing for Cycle 2 on Days 8 and 15, followed by single doses on Day 8 for Cycles 3-6. The starting dose of glofitamab for each arm may be one or more levels below the MTD/OBD determined in Part I.
  Interventions: Drug: Glofitamab; Drug: Rituximab (R); Drug: Tocilizumab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Polatuzumab vedotin

INTERVENTIONS:
Drug: Glofitamab — Glofitamab will be administered intravenously (IV) as a step-up dose for Cycle 2 on Days 8 and 15, and as a single dose from Cycle 3 onwards.
  Other Names: RO7082859
Drug: Obinutuzumab (G) — Obinutuzumab 1000 mg single dose IV infusion on Day 1 of Cycle 1 only
  Other Names: Gazyva
  Arms: Part 1: Dose Escalation r/r NHL; Part 2: DLBCL G/R-CHOP
Drug: Rituximab (R) — Rituximab will be administered as an IV infusion at a dose of 375 mg/m^2 on Day 1 of each 21-day cycle starting from Cycle 1 to Cycle 6 (Part 1) or from Cycles 1-6 (up to 8) (Part 2: DLBCL R-CHOP).
  Other Names: Rituxan
Drug: Tocilizumab — Tocilizumab will be administered as an IV infusion as per the methods described in the Summary of Product Characteristics (SmPC) or other similar local prescribing documents. Tocilizumab will be given as rescue medication.
  Other Names: Actemra
Drug: Cyclophosphamide — Cyclophosphamide 750 mg/m^2 administered IV on Day 1 of each 21-day cycle
Drug: Doxorubicin — Doxorubicin 50 mg/m^2 administered IV on Day 1 of each 21-day cycle
Drug: Vincristine — Vincristine 1.4 mg/m^2 administered by IV push on Day 1 of each 21-day cycle with a recommended cap of 2 mg
  Other Names: Oncovin
  Arms: Part 1: Dose Escalation r/r NHL; Part 2: DLBCL G/R-CHOP
Drug: Prednisone — Prednisone 100 mg/day orally on Days 1-5 (prednisone on Day 1 may be administered IV, with the remaining doses on Days 2-5 to be administered orally) of each 21-day cycle
Drug: Polatuzumab vedotin — Polatuzumab vedotin 1.8 mg/kg administered IV on Day 1 of each 21-day cycle
  Arms: Part 2: DLBCL Pola-R-CHP

SUMMARY:
This is a phase 1B, multi-center, dose-finding study of glofitamab administered in combination with obinutuzumab (Gazyva; [G]), rituximab (R) and standard doses of CHOP (G/R-CHOP or R-CHOP) in participants with r/r NHL and G/R CHOP or Pola-R-CHP in participants with untreated diffuse large B-cell lymphoma (DLBCL). Evaluating the safety, preliminary activity, pharmacokinetic (PK), and pharmacodynamic effects of this combination will be the main objectives of this study. The study is divided in two parts:

* Part I: Dose finding in participants with r/r NHL; test use of G vs R in Cycle 1
* Part II: Dose Expansion. The maximum tolerated dose or optimal biological dose (MTD or OBD) will be further assessed in participants with untreated DLBCL (>18 years of age with an age-adjusted International Prognostic Index (IPI) of 2-5). Glofitamab will be studied in combination with R-CHOP and Pola-R-CHP.

ELIGIBILITY:
Inclusion Criteria:

* Age >/=18 years
* For Part I r/r NHL dose-escalation, and Part II r/r NHL expansion: Histologically-confirmed NHL that is expected to express CD20, and which has relapsed/progressed following at least one prior treatment regimen containing R or G. Participants must be appropriate for treatment with CHOP and typically should not have been exposed to prior anthracyclines or must not exceed the cumulative lifetime dose of anthracyclines
* For Part II untreated DLBCL expansion: Histologically confirmed previously-untreated DLBCL that is expected to express CD20
* Able to provide a pretreatment biopsy between the final dose of last prior therapy and initiation of study medication at Cycle 1/Day 1
* Measurable disease, defined as at least one bi-dimensionally measurable nodal lesion, defined as >1.5 cm in its longest dimension, or at least one bi-dimensionally measurable extranodal lesion, defined as >1.0 cm in its longest dimension.
* Participants must have at least one measurable target lesion (> or = 1.5 cm) in its largest dimension by computed tomography (CT) scan
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 for participants with r/r NHL; ECOG performance status 0-3 for participants with untreated DLBCL
* Life expectancy (in the opinion of the Investigator) of 18 weeks
* Adverse events (AEs) from prior anti-cancer therapy must have resolved to Grade </= 1
* Adequate liver function
* Adequate hematological function
* Adequate renal function
* Negative serologic or polymerase chain reaction (PCR) test results for acute or chronic hepatitis B virus (HBV) infection
* Negative test results for hepatitis C virus (HCV) and human immunodeficiency virus (HIV)

Exclusion Criteria:

* Inability to comply with protocol mandated hospitalization and restrictions
* Participants with known active infection, or reactivation of a latent infection, whether bacterial, viral (including, but not limited to Epstein Barr virus (EBV), cytomegalovirus (CMV), HBV, HCV, and HIV), fungal, mycobacterial, or other pathogens (excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics (for IV antibiotics, this pertains to completion of last course of antibiotic treatment) within 4 weeks of dosing
* Prior treatment with systemic immunotherapeutic agents, including, but not limited to, radioimmuno-conjugates, antibody-drug conjugates, immune/cytokines, and monoclonal antibodies (e.g., anti-CTLA4, anti-PD1, and anti-PDL1) within 4 weeks or five half-lives of the drug, whichever is shorter, before G- or R-CHOP or Pola-R-CHP infusion on Cycle 1/Day 1
* Current Grade > 1 peripheral neuropathy by clinical examination or demyelinating form of Charcot-Marie-Tooth disease (only for participants treated in the polatuzumab vedotin arm)
* History of treatment-emergent immune-related AEs associated with prior immunotherapeutic agents, as follows: Grade >/=3 AEs, with the exception of Grade 3 endocrinopathy managed with replacement therapy; Grade 1-2 AEs that did not resolve to baseline after treatment completion
* Contraindication to any of the individual components of the immunochemotherapy
* Treatment with standard radiotherapy, any chemotherapeutic agent, or treatment with any other investigational anti-cancer agent within 4 weeks prior to study treatment at Cycle 1/Day 1 infusion
* Prior solid organ transplantation
* Prior allogeneic stem cell transplantation
* Autologous stem cell transplantation within 100 days prior to Cycle 1/Day 1
* Prior treatment with CAR T-cell therapy within 30 days prior to study treatment at Cycle 1 Day 1
* History of autoimmune disease
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* A history of confirmed progressive multifocal leukoencephalopathy
* Current or past history of central nervous system (CNS) lymphoma
* Ongoing corticosteroid use > 30 mg/day of prednisone or equivalent. Participants who received corticosteroid treatment with </=30 mg/day of prednisone or equivalent must be documented to be on a stable dose of at least 4 weeks' duration prior to Cycle 1/Day 1. Participants may have received a brief (<7 days) course of systemic steroids (</=100 mg prednisone equivalent per day) prior to initiation of study therapy for control of lymphoma-related symptoms
* Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including diabetes mellitus, history of relevant pulmonary disorders (bronchospasm, obstructive pulmonary disease), and known autoimmune diseases
* Major surgery or significant traumatic injury < 28 days prior to the study treatment infusion at Cycle 1/Day 1 (excluding biopsies) or anticipation of the need for major surgery during study treatment
* Participants with another invasive malignancy that could affect compliance with the protocol or interpretation of results
* Significant or extensive cardiovascular disease
* Left ventricular ejection fraction < 50%
* Administration of a live, attenuated vaccine within 4 weeks before study treatment infusion on Cycle 1 Day 1 or anticipation that such a live, attenuated vaccine will be required during the study
* History of illicit drug or alcohol abuse within 12 months prior to screening, in the Investigator's judgment
* Any other diseases, metabolic dysfunction, physical examination finding (including mental status), or clinical laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug
* Participants with latent or active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Part I: Percentage of Participants with Dose Limiting Toxicities (DLTs) | Up to 29 months
Part I and II: Percentage of Participants with Adverse Events | Up to 29 months

SECONDARY OUTCOMES:
Parts I and II: Percentage of Participants with a Complete Response (CR) as Assessed by the Investigator using Modified Lugano 2014 Criteria | Up to 29 months
Parts I and II: Percentage of Participants with Overall Response (Partial Response [PR] or Complete Response [CR]) | Up to 29 months
Parts I and II: Duration of Response (DOR) | Up to 29 months
Duration of CR | Up to 29 months
Progression-Free Survival (PFS) | Up to 29 months
Overall Survival (OS) | Up to 29 months
Time to First Complete Response (TFCR) | Up to 29 months
Time to First Response (TFOR) | Up to 29 months
Parts I and II: Area Under the Serum Concentration Versus Time Curve (AUC) of Glofitamab | Cycle 1 Day 1 up to 29 months
Parts I and II: Time to Maximum Serum Concentration (tmax) of Glofitamab | Cycle 1 Day 1 up to 29 months
Parts I and II: Maximum Serum Concentration (Cmax) of Glofitamab | Cycle 1 Day 1 up to 29 months
Parts I and II: Minimum Serum Concentration (Cmin) of Glofitamab | Cycle 1 Day 1 up to 29 months
Change from Baseline in T-cell Activation Markers | Up to 29 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- United States (3):
  - University of Alabama Medical Center, Birmingham, Alabama
  - Levine Cancer Institute, Charlotte, North Carolina
  - Fox Chase-Temple Cancer Center, Philadelphia, Pennsylvania
- Peter Maccallum Cancer Centre, Melbourne, Victoria, Australia
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Rigshospitalet, København Ø, Denmark
- France (3):
  - Hopital Claude Huriez, Lille
  - Hopital Hotel Dieu Et Hme, Nantes
  - Centre Henri Becquerel, Rouen
- Germany (4):
  - Universitätsklinikum Erlangen, Translational Research Center (TRC), Medizin 5, Erlangen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg, Würzburg
- Italy (4):
  - Istituto Nazionale Tumori Irccs Fondazione g. Pascale, Napoli, Campania
  - UO Ematologia, Ospedale S.Maria delle Croci, Ravenna, Emilia-Romagna
  - Asst Papa Giovanni Xxiii, Bergamo, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial, Barcelona
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, London
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham

REFERENCES:
- [Derived] Sam J, Leclercq-Cohen G, Gebhardt S, Surowka M, Herter S, Lechner K, Relf J, Briner S, Varol A, Appelt B, Domocos I, Nicolini V, Bez M, Bommer E, Jenni S, Schoenle A, Le Clech M, Colombetti S, Klein C, Umana P, Lundberg P, Korfi K, Bottos A, Bacac M. Preclinical advances in glofitamab combinations: a new frontier for non-Hodgkin lymphoma. Blood. 2025 Oct 9;146(15):1824-1836. doi: 10.1182/blood.2025028863. PMID 40749164